CLINICAL TRIAL: NCT03375034
Title: Exploring the Role of the GABAergic Modulation in Pain Transmission in Human. Effects of the GABAA Agonist N-desmethylclobazam on Central Sensitization: a Pharmacodynamic and Pharmacokinetic Study in Healthy Volunteers
Brief Title: Exploring the Role of the GABAergic Modulation in Pain Transmission in Human
Acronym: NDMC-101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jules Desmeules (Other)
Responsible Party: Sponsor-Investigator, Jules Desmeules, Prof., University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PB_2016-02140
Record Dates: First submitted 2017-09-08; First posted 2017-12-15 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Neuropathic Pain
Keywords: Chronic pain; Benzodiazepine; Central sensitization; Selective compound; GABAA receptors; Antihyperalgesia; RCT
MeSH Terms: conditions — Neuralgia; Chronic Pain | interventions — Clonazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NDMC 20mg (Experimental): oral single dose
  Interventions: Drug: NDMC 20mg
- NDMC 60mg (Experimental): oral single dose
  Interventions: Drug: NDMC60mg
- Clonazepam 1.5mg (Active Comparator): oral single dose
  Interventions: Drug: Clonazepam 1.5mg
- Placebo (Placebo Comparator): oral single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NDMC 20mg — Oral administration of one NDMC 20mg capsule and two Placebo capsules
  Arms: NDMC 20mg
Drug: NDMC60mg — Oral administration of three NDMC 20mg capsules
  Arms: NDMC 60mg
Drug: Clonazepam 1.5mg — Oral administration of three clonazepam 0.5mg capsules
  Arms: Clonazepam 1.5mg
Drug: Placebo — Oral administration of three Placebo capsules
  Arms: Placebo

SUMMARY:
Neuropathic pain affects about 7% of the general population in European countries. Meta-analyses indicate that only a minority of neuropathic pain patients has adequate response to drug therapy and management of neuropathic pain is still an unmet medical need. New insights into the contribution of defined subtypes of GABAA receptors (GABAARs) to the different clinical effects of benzodiazepines, including analgesia, have suggested that α1-sparing selective benzodiazepines, such as N-desmethylclobazam (NDMC), may be a new realistic alternative for the treatment of neuropathic pain. Results from our previous study in healthy volunteers assessing the antihyperalgesic and sedative effects of benzodiazepines on a UVB-induced pain model of central sensitization showed that, at the time of maximum effect, clobazam and clonazepam antihyperalgesic effect was greater than placebo by respectively 15.7% (95% CI 0.8 - 30.5) and 28.6% (95% CI 4.5 - 52.6), p<0.05. Moreover difference in sedation (VAS), as compared to placebo, was only significant for clonazepam 26.3mm (95%CI 15.0-37.7), p<0.001. Our preclinical data also demonstrate that, in recombinant receptors, NDMC has a better α2- over α1GABAARs activity ratio than clobazam and diazepam. And, unlike diazepam, NDMC caused no or modest sedation at antihyperalgesic doses in two strains of wild-type mice. In addition NDMC α2/α1 in vitro activity profile and long term clinical experience from its marketed parent compound (clobazam) make it an advisable clinical candidate for further proof-of-concept assessments in human. Therefore the Geneva University Hospitals have manufactured a new chemical entity and initiated a drug development program for NDMC starting with this proof-of-concept phase 1b randomized double-blind crossover (4 arms) study that will assess the analgesic and sedative effects of NDMC 20mg and 60mg compared to clonazepam 1.5 mg or placebo on a UVB-induced erythema pain model in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male subject, age between 18 and 50 years old
* Caucasian
* Type 3 skin phototype (white skin that can tan gradually and burns moderately)
* Non smoker or moderate smoker (< 10 cigarettes/day)
* No clinically abnormal findings on history and/or on physical examination
* Positive minimal erythema dose (MED) determination

Exclusion Criteria:

* Any active significant illness
* Current or past history of drug and alcohol abuse or current intake of more than 3 glasses of alcohol a day or more than 21 glasses of alcohol per week
* Psychotropic drug intake during the last month
* Sun allergy or any skin disease
* Any regular drug intake
* CYP2C19 poor metabolizer (phenotype)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Change in the area of secondary hyperalgesia from baseline | Hour 1, Hour 2, Hour 3, Hour 4, Hour 5, Hour 6, Hour 7, Hour 8, Hour 9, Hour 10 following drug administration
  The mapping of the area of secondary hyperalgesia is determined by pricking the skin surrounding the erythema with a hand-held von Frey filament (235 mN), normally felt as non-painful.
  The punctuated probe is moved along the 8 radial lines defined by the center (erythema) and the corners of a regular octagon. Testing starts outside the hyperalgesic area and the probe is moved towards the center in steps of 5 mm. The position is marked where the pin-prick sensation changes to become painful. Once complete boundaries had been defined, the areas are transcribed onto clear film and weighed. The surface area will then be calculated based on a standard measure of the weight of an area of 100cm2.

SECONDARY OUTCOMES:
Change in static mechanical pain threshold (SMPT) from baseline | Hour 1, Hour 2, Hour 3, Hour 4, Hour 5, Hour 6, Hour 7, Hour 8, Hour 9, Hour 10 following drug administration
  Increasing pressure will be manually delivered at a constant rate of 10 g / sec with a von Frey electronic device (Bioseb, Id-Tech Bioseb, Chaville, France). SMPT is defined as the lowest pressure that produces a sensation of pain. This threshold will be determined at DAY1 before UVB exposition and at DAY2 on the primary area of hyperalgesia prior to the administration of the study drug to document hyperalgesia/allodynia.
Change in dynamic mechanical sensory VAS (DMSV) from baseline | Hour 1, Hour 2, Hour 3, Hour 4, Hour 5, Hour 6, Hour 7, Hour 8, Hour 9, Hour 10 following drug administration
  Dynamic mechanical sensory is a good correlate of central sensitization and will be determined by gently stroking a hand-held cotton wool tip on the skin at a rate of approximately 1 cm/sec. Following a series of 10 strokes, the subject will be asked to score the intensity of the tactile sensation he experienced on a visual analogue scale (VAS; 0-100mm). This parameter will be determined at DAY1 before UVB exposition to document the integrity of the nociceptive fibres and at DAY2 on the primary area of hyperalgesia prior to the administration of the study drug to document hyperalgesia/allodynia.
Change in subjective feeling of sedation from baseline | Hour 1, Hour 2, Hour 3, Hour 4, Hour 5, Hour 6, Hour 7, Hour 8, Hour 9, Hour 10 following drug administration
  The subjective degree of sedation will be evaluated on a Visual Analog Scale (VAS). The subject is asked to rate on a 100 mm scale (0=not at all and100 extremely) his level of drowsiness: "How sleepy do you feel now?"
Change in memory test score from baseline | Hour 4 and Hour 10 following drug administration
  Short term anterograde memory will be tested by memorizing a list of 20 words and 30 minutes later retrieve as many of them as possible.
Change in AUC of N-desmethylclobazam from Baseline following administration of single dose (20mg, 40mg and 60mg) of N-desmethylclobazam | Hour 0.5, Hour 1, Hour 2, Hour 4, Hour 6, Hour 8, Hour 10, Hour 12, Hour 24, Hour 32, DAY 3, DAY 4, DAY 5, DAY 6, DAY 7, DAY 8, DAY 9, DAY 10, DAY 14 following drug administration
  Venous blood sample will be collected to assess N-desmethylclobazam basic pharmacokinetic parameters following single dose administration
Change in AUC of N-desmethylclobazam from Baseline following administration of repeated doses (20mg) of N-desmethylclobazam | Hour 0.5, Hour 1, Hour 2, Hour 4, Hour 6, Hour 8, Hour 10, Hour 12, Hour 24 following drug administration
  Venous blood sample will be collected to assess N-desmethylclobazam basic pharmacokinetic parameters following the administration of repeated doses of N-desmethylclobazam 20mg over 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- UGeneva, Geneva, Switzerland